CLINICAL TRIAL: NCT05140499
Title: A Prospective, Randomized Trial of Liposomal Bupivacaine Compared to Continuous Nerve Catheters on Pain Control and Post-Operative Opioid Use in Receiving Popliteal Nerve Blocks for Below the Knee Amputation
Brief Title: Liposomal Bupivacaine vs Continuous Nerve Catheters for Below the Knee Amputations
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty with enrollment
Sponsor: Aurora Quaye (Other)
Collaborators: MaineHealth (Other)
Responsible Party: Sponsor-Investigator, Aurora Quaye, Vice Chair of Research, Department of Anesthesiology and Perioperative Medicine, Maine Medical Center, MaineHealth
Organization: MaineHealth (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1807862-1
Record Dates: First submitted 2021-10-25; First posted 2021-12-01 (Actual); Results first posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Pain, Postoperative; Amputation
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single Shot Perineural Popliteal Nerve Block (Active Comparator): Single shot perineural popliteal nerve block injection of 10cc 13.3% liposomal bupivacaine combined with 15cc 0.50% bupivacaine hydrochloride within one hour prior to surgery
  Interventions: Drug: Liposomal bupivacaine
- Continuous perineural popliteal nerve block catheter (Active Comparator): Placement of continuous perineural popliteal nerve block catheter with injection of 30cc 0.5% bupivacaine within one hour prior to surgery, followed by continuous infusion of 10cc 0.3% ropivacaine (current standard practice) for at least 72 hours following surgery. Saphenous single shot 20cc 0.2
  Interventions: Drug: Bupivacaine Hydrochloride 0.5 % Injectable Solution

INTERVENTIONS:
Drug: Liposomal bupivacaine — Popliteal nerve block
  Other Names: Exparel
  Arms: Single Shot Perineural Popliteal Nerve Block
Drug: Bupivacaine Hydrochloride 0.5 % Injectable Solution — Continuous nerve catheter
  Other Names: conventional bupivacaine
  Arms: Continuous perineural popliteal nerve block catheter

SUMMARY:
Through this pilot prospective trial, we aim to obtain preliminary data investigating the effectiveness of perineural catheters and liposomal bupivacaine, both currently accepted as standard care at Maine Medical Center, for the management of post-limb amputation pain. We will use the data that we collect to inform the design of a larger, appropriately powered study.

DETAILED DESCRIPTION:
Lower extremity amputation is a common surgical procedure often due to limb ischemia or complications related to diabetes mellitus. Managing postoperative pain can be quite challenging in this patient population and persistent post-surgical pain is not uncommon. Peripheral nerve catheters (PNCs) that deliver a continuous infusion of local anesthetic have been shown to provide analgesic benefit dependent upon infusion duration and in the absence of catheter malfunction. Unfortunately, PNCs can be difficult to place and rates of dislodgement are estimated at 30%. Single shot regional nerve blocks using liposomal bupivacaine are much easier to perform than PNCs and can provide up to 72 hours of pain relief, eliminating the need for catheter placement. To date, no study has investigated the effects of liposomal bupivacaine compared to PNCs for post-surgical pain control. In this pilot study, we intend to compare pain scores, opioid consumption, and length of stay in patients randomized to both treatment strategies. We also intend to conduct an exploratory analysis investigating incidence of phantom limb pain one month following surgery. Our results will inform the design of a larger powered study to investigate treatment effects.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Physical Status Classification I-IV
* Scheduled for primary amputation or stump revision
* English speaking

Exclusion Criteria:

* Patients unable to cooperate or consent to the study
* Allergy to local anesthetics
* Existing infection at planned needle insertion site
* BMI > 40kg/m2
* Patients with a history of coagulopathy
* Emergency amputations
* Contralateral amputations
* Patients with a substance use disorder diagnosis
* Patients on opioids >90 morphine milligram equivalents (MME)/day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aurora Quaye, MD, Principal Investigator — MaineHealth
Locations (1):
- Maine Medical Center, Portland, Maine, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neil MJE. Pain after amputation. BJA Education. 2016: 16(3):107-12.
- [Background] Borg L, Howard SK, Kim TE, Steffel L, Shum C, Mariano ER. A comparison of strength for two continuous peripheral nerve block catheter dressings. Korean J Anesthesiol. 2016 Oct;69(5):506-509. doi: 10.4097/kjae.2016.69.5.506. Epub 2016 Jul 25. PMID 27703632
- [Background] Borghi B, D'Addabbo M, White PF, Gallerani P, Toccaceli L, Raffaeli W, Tognu A, Fabbri N, Mercuri M. The use of prolonged peripheral neural blockade after lower extremity amputation: the effect on symptoms associated with phantom limb syndrome. Anesth Analg. 2010 Nov;111(5):1308-15. doi: 10.1213/ANE.0b013e3181f4e848. Epub 2010 Sep 29. PMID 20881281
- [Background] Ilfeld BM. Continuous peripheral nerve blocks: a review of the published evidence. Anesth Analg. 2011 Oct;113(4):904-25. doi: 10.1213/ANE.0b013e3182285e01. Epub 2011 Aug 4. PMID 21821511
- [Background] Ilfeld BM. Continuous peripheral nerve blocks in the hospital and at home. Anesthesiol Clin. 2011 Jun;29(2):193-211. doi: 10.1016/j.anclin.2011.04.003. PMID 21620338
- [Background] Bergese SD, Ramamoorthy S, Patou G, Bramlett K, Gorfine SR, Candiotti KA. Efficacy profile of liposome bupivacaine, a novel formulation of bupivacaine for postsurgical analgesia. J Pain Res. 2012;5:107-16. doi: 10.2147/JPR.S30861. Epub 2012 May 1. PMID 22570563
- [Background] Prabhakar A, Ward CT, Watson M, Sanford J, Fiza B, Moll V, Kaye RJ, Morgan Hall O, Cornett EM, Urman RD, Kaye AD. Liposomal bupivacaine and novel local anesthetic formulations. Best Pract Res Clin Anaesthesiol. 2019 Dec;33(4):425-432. doi: 10.1016/j.bpa.2019.07.012. Epub 2019 Jul 19. PMID 31791561
- [Background] Davidovitch R, Goch A, Driesman A, Konda S, Pean C, Egol K. The Use of Liposomal Bupivacaine Administered With Standard Bupivacaine in Ankle Fractures Requiring Open Reduction Internal Fixation: A Single-Blinded Randomized Controlled Trial. J Orthop Trauma. 2017 Aug;31(8):434-439. doi: 10.1097/BOT.0000000000000862. PMID 28430722
- [Background] Mazloomdoost D, Pauls RN, Hennen EN, Yeung JY, Smith BC, Kleeman SD, Crisp CC. Liposomal bupivacaine decreases pain following retropubic sling placement: a randomized placebo-controlled trial. Am J Obstet Gynecol. 2017 Nov;217(5):598.e1-598.e11. doi: 10.1016/j.ajog.2017.07.001. Epub 2017 Jul 8. PMID 28694151
- [Background] Yan Z, Chen Z, Ma C. Liposomal bupivacaine versus interscalene nerve block for pain control after shoulder arthroplasty: A meta-analysis. Medicine (Baltimore). 2017 Jul;96(27):e7226. doi: 10.1097/MD.0000000000007226. PMID 28682872
- [Background] Hussain N, Brull R, Sheehy B, Essandoh MK, Stahl DL, Weaver TE, Abdallah FW. Perineural Liposomal Bupivacaine Is Not Superior to Nonliposomal Bupivacaine for Peripheral Nerve Block Analgesia. Anesthesiology. 2021 Feb 1;134(2):147-164. doi: 10.1097/ALN.0000000000003651. PMID 33372953
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Background] Richardson C, Glenn S, Nurmikko T, Horgan M. Incidence of phantom phenomena including phantom limb pain 6 months after major lower limb amputation in patients with peripheral vascular disease. Clin J Pain. 2006 May;22(4):353-8. doi: 10.1097/01.ajp.0000177793.01415.bd. PMID 16691088
- [Background] Jensen TS, Krebs B, Nielsen J, Rasmussen P. Immediate and long-term phantom limb pain in amputees: incidence, clinical characteristics and relationship to pre-amputation limb pain. Pain. 1985 Mar;21(3):267-278. doi: 10.1016/0304-3959(85)90090-9. PMID 3991231
- [Background] Madabhushi L, Reuben SS, Steinberg RB, Adesioye J. The efficacy of postoperative perineural infusion of bupivacaine and clonidine after lower extremity amputation in preventing phantom limb and stump pain. J Clin Anesth. 2007 May;19(3):226-9. doi: 10.1016/j.jclinane.2006.07.008. PMID 17531734
- [Background] Jahangiri M, Jayatunga AP, Bradley JW, Dark CH. Prevention of phantom pain after major lower limb amputation by epidural infusion of diamorphine, clonidine and bupivacaine. Ann R Coll Surg Engl. 1994 Sep;76(5):324-6. PMID 7979074
- [Background] Lambert Aw, Dashfield Ak, Cosgrove C, Wilkins Dc, Walker Aj, Ashley S. Randomized prospective study comparing preoperative epidural and intraoperative perineural analgesia for the prevention of postoperative stump and phantom limb pain following major amputation. Reg Anesth Pain Med. 2001 Jul-Aug;26(4):316-21. doi: 10.1053/rapm.2001.23934. PMID 11464349
- [Background] Nikolajsen L, Ilkjaer S, Christensen JH, Kroner K, Jensen TS. Randomised trial of epidural bupivacaine and morphine in prevention of stump and phantom pain in lower-limb amputation. Lancet. 1997 Nov 8;350(9088):1353-7. doi: 10.1016/S0140-6736(97)06315-0. PMID 9365449
- [Background] Nikolajsen L, Ilkjaer S, Jensen TS. Effect of preoperative extradural bupivacaine and morphine on stump sensation in lower limb amputees. Br J Anaesth. 1998 Sep;81(3):348-54. doi: 10.1093/bja/81.3.348. PMID 9861117
- [Background] Morey TE, Giannoni J, Duncan E, Scarborough MT, Enneking FK. Nerve sheath catheter analgesia after amputation. Clin Orthop Relat Res. 2002 Apr;(397):281-9. doi: 10.1097/00003086-200204000-00032. PMID 11953619
- [Background] Dworkin RH, Turk DC, Revicki DA, Harding G, Coyne KS, Peirce-Sandner S, Bhagwat D, Everton D, Burke LB, Cowan P, Farrar JT, Hertz S, Max MB, Rappaport BA, Melzack R. Development and initial validation of an expanded and revised version of the Short-form McGill Pain Questionnaire (SF-MPQ-2). Pain. 2009 Jul;144(1-2):35-42. doi: 10.1016/j.pain.2009.02.007. Epub 2009 Apr 7. PMID 19356853
- [Background] Gallagher P, MacLachlan M. Development and psychometric evaluation of the Trinity Amputation and Prosthesis Experience Scales (TAPES). Rehabilitation Psychology. 2000: 45(2), 130-154.
- [Background] Jensen MP, Castarlenas E, Tome-Pires C, de la Vega R, Sanchez-Rodriguez E, Miro J. The Number of Ratings Needed for Valid Pain Assessment in Clinical Trials: Replication and Extension. Pain Med. 2015 Sep;16(9):1764-72. doi: 10.1111/pme.12823. Epub 2015 Jul 14. PMID 26178637
- [Background] Julious SA. Sample size of 12 per group rule of thumb for a pilot study. Pharmaceutical Statistics. 2005;4(4):287-91.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Shot Perineural Popliteal Nerve Block | Continuous Perineural Popliteal Nerve Block Catheter
Started | 5 | 6
Completed | 4 | 4
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Shot Perineural Popliteal Nerve Block | Continuous Perineural Popliteal Nerve Block Catheter | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (10.1) | 52.0 (18.6) | 54 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 6 | 11
  Unknown or Not Reported | 0 | 0 | 0
Daily Opioid Use [Median (Full Range); unit: MME/day] — Daily opioid dose (in MME) prior to surgery, for participants taking opioids Population: The analysis only includes participants who were taking a daily opioid prior to surgery.
  MME/day
    number analyzed (Participants) | 2 | 3 | 5
    (all) | 22.5 [15 to 30] | 40 [30 to 40] | 30 [15 to 40]

OUTCOME MEASURES:

1. Primary Outcome: Pain Assessed by Numerical Rating Scale (NRS)
Description: Average NRS pain scores (0-10, 0=no pain, 10=worst possible pain)
Time Frame: 72 hours post-operatively
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Single Shot Perineural Popliteal Nerve Block | Continuous Perineural Popliteal Nerve Block Catheter
Number analyzed (Participants) | 5 | 6
score on a scale | 6 (3.07) | 4 (3.32)

2. Secondary Outcome: Opioid Consumption
Description: Total amount of opioid medication given, in morphine milligram equivalents
Time Frame: 72 hours post-operatively
Measure: Median (Inter-Quartile Range); unit: MME
Arm/Group | Single Shot Perineural Popliteal Nerve Block | Continuous Perineural Popliteal Nerve Block Catheter
Number analyzed (Participants) | 5 | 6
MME | 151 [85 to 330] | 47 [15 to 231]

3. Secondary Outcome: Post-operative Length of Stay
Description: Post-operative length of stay in hours
Time Frame: Measured from surgical stop time to discharge time, an average of 5 days.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Single Shot Perineural Popliteal Nerve Block | Continuous Perineural Popliteal Nerve Block Catheter
Number analyzed (Participants) | 5 | 6
hours | 121.9 [89.0 to 145.0] | 118.3 [96.9 to 340.8]

4. Secondary Outcome: Post-operative Pain Assessed by the Short Form McGill Pain Questionnaire-2 (SFMPQ-2)
Description: Total SFMPQ-2 score (low score of 0, no pain to a high score of 220, worst possible pain)
Time Frame: 30 days following surgery
Population: 3 participants overall were lost to follow-up
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Single Shot Perineural Popliteal Nerve Block | Continuous Perineural Popliteal Nerve Block Catheter
Number analyzed (Participants) | 4 | 4
units on a scale | 14 [0 to 35] | 13 [0 to 43]

5. Secondary Outcome: Phantom Limb Pain Assessed Using Questions From the Trinity Amputation and Prosthesis Experiences Scales-Revised (TAPES-R)
Description: Phantom Limb Pain was measured using questions 4 and 5 from Part II of the TAPES-R (scores can range from 0, no pain, to 22, severe pain)
Time Frame: 30 days following surgery
Population: 3 participants overall were lost to follow-up
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Single Shot Perineural Popliteal Nerve Block | Continuous Perineural Popliteal Nerve Block Catheter
Number analyzed (Participants) | 4 | 4
units on a scale | 0.25 [0 to 1] | 0.75 [0 to 3]

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Single Shot Perineural Popliteal Nerve Block | Continuous Perineural Popliteal Nerve Block Catheter
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 0/5 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT05140499/Prot_SAP_000.pdf